CLINICAL TRIAL: NCT07260669
Title: A Phase 2, Randomized, Double-blind, Placebo-controlled Trial to Investigate the Efficacy and Safety of 2 Doses of Vipoglanstat in Patients With Moderate to Severe Endometriosis-related Pain - the NOVA Trial
Brief Title: A Phase 2 Trial to Investigate Efficacy and Safety of Vipoglanstat in Women With Endometriosis
Acronym: NOVA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Gesynta Pharma AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GS-248-203; 2025-522452-16-00 (EU CTIS Number)
Record Dates: First submitted 2025-09-29; First posted 2025-12-03 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Endometriosis
Keywords: Non-menstrual pelvic pain; Dysmenorrhea; Pelvic pain
MeSH Terms: conditions — Endometriosis; Dysmenorrhea; Pelvic Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dose A Vipoglanstat (Experimental)
  Interventions: Drug: Vipoglanstat
- Dose B Vipoglanstat (Experimental)
  Interventions: Drug: Vipoglanstat
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vipoglanstat — Participants will receive vipoglanstat capsules orally for approximately 4 menstrual cycles during the treatment period.
  Arms: Dose A Vipoglanstat; Dose B Vipoglanstat
Drug: Placebo — Participants will receive matching placebo capsules orally for approximately 4 menstrual cycles during the treatment period.
  Arms: Placebo

SUMMARY:
The main objective of the trial is to evaluate the efficacy of vipoglanstat on endometriosis-related non-menstrual pelvic pain (NMPP).

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal females 18 to < 45 years of age at the time of Visit 1.
* Endometriosis diagnosis confirmed and documented within the last 10 years prior to Visit 1 or during Visit based on:

  * Surgical (via direct visualization or biopsy verified) or
  * Imaging (ie, endometriotic lesion(s) detected by transvaginal sonography or magnetic resonance imaging [MRI].
* History of NMPP significantly affecting daily life confirmed at Visit 1.
* The participant reports moderate, severe, or very severe pain during non-menstrual days in the month prior to Visit 2, based on patient global assessment NMPP.

Exclusion Criteria:

* Chronic pelvic pain that is not judged to be primarily related to endometriosis (eg, chronic pelvic infection, interstitial cystitis, nerve entrapments or neuropathies, non-endometriosis-related pelvic adhesive disease, persistent symptomatic ovarian cyst [eg, dermoid], posttubal ligation, symptomatic hydrosalpinx, and vaginismus).
* Has had more than 2 surgical procedures for endometriosis.

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 190 (Estimated)
Dates: Start 2025-10-15 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants who meet the Predefined NMPP Responder Criteria from Baseline to Fourth Month of Treatment | Baseline to 4 months

SECONDARY OUTCOMES:
Change in Mean Worst NMPP numeric Rating Scale (NRS) Score from Baseline to Fourth Month of Treatment | Baseline to 4 months
Percentage of Participants who Meet the Predefined Dysmenorrhea Responder Criteria from Baseline to Fourth Month of Treatment | Baseline to 4 months
Change in Mean Worst Dysmenorrhea NRS Score from Baseline to Fourth Month of Treatment | Baseline to 4 months
Change in Endometriosis Health Profile 30 Item Patient Reported Outcome (EHP-30) Score from Baseline to End of Treatment | Baseline to 4 months
Change in EHP-30 Sexual Intercourse Subscale Score from Baseline to End of Treatment | Baseline to 4 months
Change in Mean Daily Opioid Rescue Medication Use for NMPP from Baseline to Fourth Month of Treatment | Baseline to 4 months
Change in Mean Daily Opioid Rescue Medication Use for Dysmenorrhea from Baseline to Fourth Month of Treatment | Baseline to 4 months
Number of Participants with Adverse Events | Up to 10 months
  Any clinically significant changes in laboratory variables, including clinical chemistry, hematology, and urinalysis will be reported as adverse events.

CONTACTS AND LOCATIONS:
Locations (26):
- Bulgaria (2):
  - MHAT Puls AD, Blagoevgrad
  - Lyulin Hospital, Sofia
- Czechia (3):
  - Gynekologie MEDA s.r.o, Brno
  - NEUMED Gynekologicka Ambulance s.r.o., Olomouc
  - STELLA-GYN, s.r.o., Vodňany
- Hungary (4):
  - MedEnd, Budapest
  - Robert Karoly Private Hospital Tritonlife Medical Center, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Somogy Varmegyei Kaposi Mor Oktato Korhaz (Kaposi Mor County Hospital), Kaposvár
- Poland (10):
  - Prywatna Klinika Polozniczo - Ginekologiczna Sp. Z O.O., Bialystok
  - NZOZ Medem, Katowice
  - Centrum Medyczne Angelius Provita, Katowice
  - NZOZ Vita Longa Sp. z o.o., Katowice
  - Medico Praktyka Lekarska, Krakow
  - Centrum Medyczne Chodzki, Lublin
  - ETG Siedlce, Siedlce
  - Aidport sp. Z o.o., Skorzewo
  - Twoja Przychodnia SCM, Szczecin
  - Specjalistyczna Praktyka Lekarska Krzysztof Dynowski, Warsaw
- United Kingdom (7):
  - Accellacare Yorkshire, Bradford
  - Accellacare Northamptonshire, Corby
  - Accellacare Warwickshire, Coventry
  - Accellacare North London, Northwood
  - Norfolk and Norwich University Hospital - Norfolk and Norwich University Hospitals NHS Foundation Trust, Norwich
  - Accellacare South London, Orpington
  - University of Oxford, Oxford

IPD SHARING:
Plan to Share IPD: No